CLINICAL TRIAL: NCT03740594
Title: Effect of Kangaroo Mother Care and Its Duration on Neurobehavioral Performance and Stress Response of Preterm Neonates
Brief Title: Effect of KMC on Neurobehavior of Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Mohamed Mohamed Shinkar, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Effect of KMC on neurobehavior
Record Dates: First submitted 2018-11-10; First posted 2018-11-14 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Neonatal Neurobehavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KMC 60 min group (Active Comparator)
  Interventions: Behavioral: KMC
- KMC 120 min group (Active Comparator)
  Interventions: Behavioral: KMC
- control group (Active Comparator)
  Interventions: Behavioral: KMC

INTERVENTIONS:
Behavioral: KMC — Neonates were subjected to either daily KMC for 60 minutes, daily KMC for 120 minutes or conventional care (controls) for at least 7 days.

SUMMARY:
This prospective cohort study was conducted on stable preterm infants (31 to 35 weeks gestation). Neonates were subjected to either daily KMC for 60 minutes, daily KMC for 120 minutes or conventional care (controls) for at least 7 days. Neonates were evaluated by Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS) at 36 weeks gestation. Salivary cortisol was measured before and after first KMC session and after 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Stable preterm neonates with gestational age between 31 and 35 weeks.

Exclusion Criteria:

* Neonates with major congenital birth defects or chromosomal anomalies.
* Perinatal asphyxia and intra-ventricular hemorrhage.
* Hemodynamically significant cardiac abnormalities.
* Neonates received postnatal steroids.
* Neonates whose mothers had a history of drug abuse during pregnancy.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS) | the age of 36 weeks
  applying Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS) which is used to assess the neuro-behavioral performance of neonates.It consists of 13 subscales :Habituation, Attention, Arousal, Regulation, Handling procedures, Quality of movement, Excitability, Lethargy, Non-optimal reflexes, Asymmetric reflexes, Hypertonicity, and Stress/abstinence scale.Scores of subscales are from 1 to 9.
Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS) | the age of 36 weeks
  applying Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS) which is used to assess the neuro-behavioral performance of neonates.It consists of 13 subscales :Habituation, Attention, Arousal, Regulation, Handling procedures, Quality of movement, Excitability, Lethargy, Non-optimal reflexes, Asymmetric reflexes, Hypertonicity, and Stress/abstinence scale.Scores of subscales are from 1 to 9. For stress, lethargy, non-optimal response and asymmetic reflexes, the higher the seb-scale, the worse. In other sub-scales, the higher the scale, the better.

SECONDARY OUTCOMES:
Salivary cortisol | 7 days
  measuring salivary cortisol

IPD SHARING:
Plan to Share IPD: No